CLINICAL TRIAL: NCT01983891
Title: Improving Nutritional Outcomes Among Food Insecure Twin Cities Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013NTLS011
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Change in Dietary Outcomes
Keywords: food shelf; nutrition education; cooking course

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): 6-week nutrition education and cooking course
  Interventions: Other: Cooking course

INTERVENTIONS:
Other: Cooking course — 6-week nutrition education and cooking course

SUMMARY:
This is a pilot intervention study conducted in four food shelves in the Twin Cities area. The aims of the study are to improve nutritional outcomes and client skills and self-efficacy among a culturally diverse group of food shelf clients through a nutrition education and meal preparation program. This study will also identify opportunities to expand the supply of healthy and culturally relevant foods in food shelves. The goal is to inform a larger-scale intervention to improve the nutritional quality and cultural relevance of food shelf items as well as client outcomes. The primary outcome is participant change in Health Eating Index scores from pre-intervention to post-intervetion.

DETAILED DESCRIPTION:
Food insecurity disproportionately affects low-income, minority, and foreign-born families, resulting in a disproportionate burden of nutrition-related chronic conditions affecting these groups. In Minnesota, over a half a million food insecure families relied on food shelves (also known as food pantries) for emergency food assistance in 2009. Yet reliance on food shelves in a culturally diverse population may present nutritional challenges for two main reasons. First, unlike many food assistance programs (e.g., school nutritional programs, WIC), there are currently no existing standards on the nutritional quality of food shelf offerings. Inventory data collected from a sample of Twin Cities food shelves in the summer of 2012 began to identity priority areas for the improvement of the nutritional quality of food shelves items, but such recommendations have yet to be implemented. Second, securing healthy meals for the large population of immigrants and refugees families who rely on food shelves in the Twin Cities may be particularly challenging. Among these clients, unfamiliarity with "American" foods and cooking practices for foods that are most affordable or available may serve as barriers to healthy meal preparation. Very little research has examined the potential for cooking skills and the incorporation of new foods in improving dietary outcomes among a group of culturally diverse food insecure families.

Recognizing that nutritional outcomes are driven by influence at both the food systems level and the individual level, the long-term goal of this research is to improve nutritional outcomes among food insecure families through enhancements at both the food shelf level and the client level. Because of the complexity in making systemic improvements in the quality of the emergency food supply, this pilot study will conduct formative research on improving food supply at the food shelf level, while primarily focusing on testing strategies to improve nutrition-related behaviors at the client level.

This intervention will focus primarily on promoting cooking skills using healthier "American" items along with culturally appropriate ingredients. Cooking classes will occur through a partnership with the Cooking Matters™ program, which leads hands-on 6-week cooking based nutrition education programs at a variety of venues in the greater Twin Cities area, and is conducted by the University of Minnesota Extension.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 18 and older
* Required food assistance from a participating food shelf in the last 30 days
* Must be willing to give verbal consent

Exclusion Criteria:

* Not able to speak and understand English
* Potential participants who have an apparent or self-reported physical or mental disability that would prohibit them from participating in a cooking course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Healthy Eating Index score | 3 months
  The Healthy Eating Index is scored on a scale of 0 to 100 and will be analyzed as a continuous outcome. Mean change in index score T1 to T2 will be assessed using a paired t-test with each individual serving as his or her own control.

SECONDARY OUTCOMES:
Meal preparations skills and self-efficacy | 3 months
  Meal preparation skills and self-efficacy will be measured by 10 Likert scale items.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Caspi, ScD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Department of Family Medicine and Community Health, Minneapolis, Minnesota, United States